CLINICAL TRIAL: NCT03661866
Title: A Longitudinal Observational Study of Patients Undergoing Therapy for Immune-Mediated Inflammatory Skin Conditions
Brief Title: A Longitudinal Observational Study of Patients Undergoing Therapy for IMISC
Acronym: TARGET-DERM
Status: Recruiting | Type: Observational
Sponsor: Target PharmaSolutions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TARGET-DERM
Record Dates: First submitted 2018-09-04; First posted 2018-09-07 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-05

CONDITIONS: Atopic Dermatitis; Alopecia Areata; Hidradenitis Suppurativa; Vitiligo; Psoriasis; Chronic Spontaneous Urticaria
Keywords: Atopic Dermatitis; IMISC; Registry; Observational; Immune-mediated Inflammatory Skin Conditions
MeSH Terms: conditions — Dermatitis, Atopic; Alopecia Areata; Hidradenitis Suppurativa; Vitiligo; Psoriasis; Chronic Urticaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Biospecimen Retention: Samples With DNA — Patients enrolled in TARGET-DERM may be invited to participate in the Biorepository Bank (BSB). Blood, buccal and tape strip samples for biomarker and DNA assays will be collected on a voluntary basis and participation in this project will not affect participation in the main study. These samples will be shipped to a central repository for storage to use in future studies. Samples stored at the biorepository will be identified only with the participant's unique study identification (ID) number and the date the sample was obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
TARGET-DERM is a longitudinal, observational study of adult and pediatric patients being managed for Atopic Dermatitis and other Immune-Mediated Inflammatory Skin Conditions (IMISC) in usual clinical practice. TARGET-DERM will create a research registry of patients with IMISC within academic and community real-world practices in order to assess the safety and effectiveness of current and future therapies.

DETAILED DESCRIPTION:
TARGET-DERM is a longitudinal, observational study of adult and pediatric patients being managed for Atopic Dermatitis and other Immune-Mediated Inflammatory Skin Conditions (IMISC) in usual clinical practice. TARGET-DERM will create a research registry of patients with IMISC within academic and community real-world practices in order to assess the safety and effectiveness of current and future therapies.

The duration of follow-up for participants enrolled in the EU is limited to 5-years. Those within in US and Canada may consent to indefinite follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults and children (all ages) with Atopic Dermatitis or other Immune-mediated Inflammatory Skin Conditions been prescribed any dermatologic treatment.
* 2. Participant has plans for future visits at the site for continued management of IMISC.

Exclusion Criteria:

* 1. Inability to provide written informed consent/assent.
* 2. Subjects participating in any interventional study or trial for IMISC treatment trial at the time of enrollment. Patients may be enrolled in TARGET-DERM once participation in the trial is complete. Note: Participants may be enrolled in other registries or studies where IMISC treatment outcomes are observed and/or reported (such as center-based registries).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children (all ages) with with Atopic Dermatitis or other IMISC been prescribed any dermatologic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2018-12-21 (Actual); Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Characterize IMISC Treatment Regimens in Clinical Practice | 25 Years
  Enable characterization of IMISC disease activity and comorbid medical conditions over time.
Evaluate Patient Outcomes in Clinical Practice | 25 Years
  Enable characterization of IMISC disease activity and comorbid medical conditions over time.
Evaluate Adverse Events of IMISC and treatment in Clinical Practice | 25 Years
  Enable characterization of IMISC disease activity and comorbid medical conditions over time.

SECONDARY OUTCOMES:
Evaluate the relationship between IMISC and comorbid medical conditions | 25 Years
  Inform clinical practice by identifying the occurrence and impact of comorbid medical conditions on treatment regimens, utilize patient reported outcomes, and evaluate patient support programs.
Evaluate Patient Reported Outcome (PRO) measures | 25 Years
  Inform clinical practice by identifying the occurrence and impact of comorbid medical conditions on treatment regimens, utilize patient reported outcomes, and evaluate patient support programs.
Evaluate outcomes related to Patient Support Programs (PSPs) | 25 Years
  Inform clinical practice by identifying the occurrence and impact of comorbid medical conditions on treatment regimens, utilize patient reported outcomes, and evaluate patient support programs.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dalfonso, Study Director — Target RWE
Locations (63):
- United States (54):
  - Clear Dermatology & Aesthetics Center/Investigative MD, Scottsdale, Arizona
  - Johnson Dermatology, Fort Smith, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Arkansas Dermatology, Little Rock, Arkansas
  - First OC Dermatology, Fountain Valley, California
  - Center for Dermatology Cosmetic and Laser Surgery, Fremont, California
  - University of California, Irvine, California
  - University of California - San Diego/Rady Children's Hospital, San Diego, California
  - George Washington University, Washington D.C., District of Columbia
  - Feinstein Dermatology and Cosmetic Surgery, Hollywood, Florida
  - Academic Alliance in Dermatology, Tampa, Florida
  - Integrated Dermatology of West Palm Beach, West Palm Beach, Florida
  - Lurie Children's Hospital/Northwestern University, Chicago, Illinois
  - Dawes Fretzin Dermatology/ Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Family Allergy and Asthma Research Institute, Louisville, Kentucky
  - DermAssociates, LCC, Rockville, Maryland
  - Integrated Dermatology of Massachusetts, Quincy, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Carl Thornblade, MD, PLLC, Missoula, Montana
  - South Lincoln Dermatology Clinic, Lincoln, Nebraska
  - Advanced Dermatology of the Midlands, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Windsor Dermatology, East Windsor, New Jersey
  - Linda Susan Marcus, Wyckoff, New Jersey
  - Centurion Dermatology, Brooklyn, New York
  - The University of Buffalo, Buffalo, New York
  - Empire Dermatology, East Syracuse, New York
  - Forest Hills Dermatology Group, Forest Hills, New York
  - Greenwich Village Dermatology, New York, New York
  - Ichan School of Medicine, New York, New York
  - Advanced Allergy & Asthma, PLLC, Rockville Centre, New York
  - Montefiore Medical Center, The Bronx, New York
  - Allergy Partners of Western North Carolina, Asheville, North Carolina
  - UNC Dermatology, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Allergy and Clinical Immunology, Pittsburgh, Pennsylvania
  - The Medical University of South Carolina, Charleston, South Carolina
  - El Paso Dermatology Center, El Paso, Texas
  - North Texas Center for Clinical Research, Frisco, Texas
  - Asthma and Allergy Center, Lewisville, Texas
  - Center for Clinical Studies, Webster, Texas
  - Allergy Associates of Utah, Murray, Utah
  - University of Utah MidValley Dermatology, Murray, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - North Sound Dermatology, Mill Creek, Washington
  - Spokane Dermatology Clinic, Spokane, Washington
  - Dermatology Center for Skin Health, Morgantown, West Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (4):
  - Skin Centre for Dermatology, Peterborough, Ontario
  - York Dermatology Clinic and Research Centre, Richmond Hill, Ontario
  - Innovaderm Research, Inc., Montreal, Quebec
  - Saskatoon Dermatology Centre, Saskatoon, Saskatchewan
- Germany (3):
  - Dermatologische Gemeinschaftspraxis Mahlow, Mahlow, Bradenburg
  - Dr. Bernhard Korge, Düren, North Rhine-Westphalia
  - UKSH- Institut für Entzündungsmedizin, Lübeck, Schleswig-Holstein
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario La Princesa, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abuabara K, Silverberg JI, Simpson EL, Paller AS, Eichenfield LF, Bissonnette R, Krueger J, Harris JE, Dalfonso L, Watkins SE, Crawford JM, Thaci D, Guttman-Yassky E. International observational atopic dermatitis cohort to follow natural history and treatment course: TARGET-DERM AD study design and rationale. BMJ Open. 2020 Nov 27;10(11):e039928. doi: 10.1136/bmjopen-2020-039928. PMID 33247014